CLINICAL TRIAL: NCT01351233
Title: Evaluation of the Rotational Stability of The AcrySof Toric Intraocular Lens in the Capsular Bag in High Myopic Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, A-Yong Yu, Wenzhou Medical College, Ayong Yu MD,PhD Eye Hospital, Wenzhou Medical College, China., Wenzhou Medical University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: WMC
Record Dates: First submitted 2011-05-06; First posted 2011-05-10 (Estimated); Last update posted 2012-07-06 (Estimated); Status verified 2012-07

CONDITIONS: Cataract
Keywords: Cataract
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Cataract Surgery — Take the operation of phacoemulsification and implant the AcrySof Toric intraocular lens into the capsular bag in high myopic subjects.
  Other Names: refractive lens exchange surgery

SUMMARY:
The purpose of this study is to evaluate the stability and efficacy of The AcrySof Toric intraocular lens in the bag in high myopic subjects.

DETAILED DESCRIPTION:
According to numerous estimations, 15% to 29% of patients with cataract have≥1.5 diopters (D) of refractive astigmatism. New toric IOL designs (Acrysof © toric IOL; Alcon), approved by the US Food and Drug Administration (FDA) at the end of 2005, have been found to be more stable and safety in the capsular bag in subjects with normal axis length of eye. Then,this study aims at the confirmation of the stability of The AcrySof Toric intraocular lens in the bag in high myopic subjects.Then we may find a more effective treatment for the high myopic patients with complicated cataract and sever cornea astigmatism .

ELIGIBILITY:
Inclusion Criteria:

1. Sphere more than -6.0D;
2. Cornea astigmatism from -1.0 D to -4.0D;
3. Clinical diagnosis of complicated cataract;
4. Ask for and accept refractive lens exchange surgery;
5. Accept AcrySof Toric intraocular lens .

Exclusion Criteria:

1. Other eye diseases induces impaired vision ,such as retinal detachment,keratoconus,pterygium,glaucoma,choroidal detachment,vitreous hemorrhage,congenital cataract,lens dislocation,anterior uveitis ,pupil deformation and so on;
2. Previous corneal or intraocular surgery;
3. Refuse surgery;
4. Refuse to use AcrySof Toric intraocular lens .

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
The position of IOL | 6 months
  Postoperatively, with the patient sitting upright,the position of IOL was assessed by slit lamp。Then ，We would calculate the rotation of IOL .

SECONDARY OUTCOMES:
refraction astigmatism | 6 months
  We would like to evaluate the improvement of refraction astigmatism after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ayong Yu, Ph.D., Study Director — Wenzhou Medical University
Locations (1):
- Wenzhou Medical College, Wenzhou, Zhejiang, China